CLINICAL TRIAL: NCT03234465
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Topically-applied AG013 for the Attenuation of Oral Mucositis in Subjects With Cancers of the Head and Neck Receiving Concomitant Chemoradiation Therapy
Brief Title: Efficacy, Safety and Tolerability of AG013 in Oral Mucositis Compared to Placebo When Administered Three Times Per Day
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No efficacy could be demonstrated, sponsor decided to prematurely end the study.
Sponsor: Oragenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG013-ODOM-201
Record Dates: First submitted 2017-07-21; First posted 2017-07-31 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG013: three mouth rinses/day (Experimental): Subjects will rinse three times per day with AG013 mouth rinse beginning from the start of radiotherapy until 2 weeks following its completion. The active treatment phase lasts for 7 to 9 weeks, depending on the duration of radiotherapy.
  Interventions: Biological: AG013
- Placebo: three mouth rinses/day (Placebo Comparator): Subjects will rinse three times per day with placebo mouth rinse beginning from the start of radiotherapy until 2 weeks following its completion. The active treatment phase lasts for 7 to 9 weeks, depending on the duration of radiotherapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AG013 — AG013 is made up of genetically modified (GM) bacteria called Lactococcus lactis (L. lactis). Wild type L. lactis are commonly used to produce dairy products including cheeses and milk. To make AG013, the DNA of L. lactis has been changed in the laboratory to secrete a protein called human Trefoil Factor 1 (hTFF1). hTFF1 is normally secreted in saliva and intestines. Trefoil factors have been shown to be important in protecting and healing mucosal tissues, such as the tissue in the mouth, when these tissues are damaged by cancer therapies such as chemotherapy and radiation therapy.
  Arms: AG013: three mouth rinses/day
Other: Placebo — Subjects assigned to the placebo group will receive appearance- and taste-matched placebo powder.
  Arms: Placebo: three mouth rinses/day

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety and tolerability of topically administered AG013 compared to placebo for reducing Oral Mucositis (OM) in patients undergoing chemoradiation for the treatment of head and neck cancer, as measured by the duration, time to development, and overall incidence of OM during the active treatment phase, beginning from the start of chemoradiation therapy (CRT) until 2 weeks following its completion.

The effect of AG013 on patient-reported symptoms and analgesic use during the active treatment phase, and on the cumulative radiation dose administered before the onset of OM will also be evaluated, as will biomarkers and, in a subset of subjects, the PK (pharmacokinetic) profile of AG013.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, placebo-controlled, 2-arm, multi-center trial in which subjects will be randomized in a 1:1 ratio to receive either placebo or AG013. AG013 is a mouth rinse formulation of Lactococcus lactis strain sAGX0085, deficient in the gene coding for thymidylate synthase and producing human TFF1 (Trefoil Factor 1).

Approximately 200 subjects will be enrolled in the study. To protect subjects from unanticipated safety risks, enrollment and treatment in the double-blind study will continue until 10 subjects on AG013 have been recruited. The Data Safety Monitoring Board (DSMB) will review safety data after these 10 subjects on AG013 have completed study treatment. If there are no safety signals identified, the study will continue to recruit the planned number of subjects.

There are 4 study periods as described below: screening, active treatment, short term follow-up and long term follow-up. The screening phase will be no longer than 4 weeks. The active treatment phase will be between 7 and 9 weeks depending on the subject's prescribed CRT (chemoradiation therapy) plan. The short term follow-up phase will be 4 weeks in duration. The long term follow-up will continue until 12 months post CRT. Oral mucositis (OM) assessments will begin at the start of CRT and continue until the subject has completed short term follow-up or until the OM resolves (as defined by a WHO (World Health Organization) score of ≤ 1), whichever comes first. Long term follow-up will continue for 12 months to assure that AG013 does not adversely impact the tumor response to anti-neoplastic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign the study specific Informed Consent Form
2. Pathologically-confirmed squamous cell carcinoma of the oral cavity, oropharynx, nasopharynx or hypopharynx or HPV-positive unknown primaries presumed to be of oropharyngeal, nasopharyngeal or hypopharyngeal origin
3. Tumor HPV status established
4. Planned to receive either primary or post-operative CRT
5. Planned IMRT (Intensity-Modulated Radiotherapy)
6. Planned administration of cisplatin administered weekly or tri-weekly during RT
7. Males or females 21 years or older
8. Karnofsky performance score (KPS) ≥ 70%
9. Screening laboratory assessments:

   * Hemoglobin ≥ 10g/dl
   * White blood count ≥ 3500 cells/mm3
   * Absolute neutrophil counts ≥ 1500 cells/ mm3
   * Serum AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤ 3 x ULN
   * Calculated Creatinine Clearance ≥ 50 ml/min
   * Negative pregnancy test (serum or urine) for females of childbearing potential performed 7 days before IMP (Investigational Medicinal Product) administration.
10. Subjects of childbearing potential must confirm to use an effective method of birth control during study participation and for 30 days following the last treatment with IMP. Male subjects, when having hetero-sexual intercourse with a female of childbearing potential must use a condom during study participation and 90 days following the last treatment with IMP and their partner should use an effective method of birth control during that period as well.

Exclusion Criteria:

1. Prior radiation to the head and neck
2. Increased risk of developing infectious endocarditis
3. Prior gene therapy
4. Presence of active infectious oral disease
5. Presence of any oral lesions that may confound the ability to assess oral mucositis grade
6. Current use of antibiotic rinses or troches
7. Herbal, alternative remedies, and alcohol containing over-the-counter mouthwashes are excluded during the course of the study
8. Current alcohol abuse syndrome
9. Chronic immunosuppression
10. Known seropositive for HIV
11. Use of investigational agent within 30 days of signing informed consent
12. Tooth extraction prior to radiation in which the extraction site is not epithelialized
13. Signs and symptoms of active dental disease
14. Female subjects who are pregnant or nursing
15. Known allergy to excipients of the IMP
16. Inability to give informed consent or comply with study requirements
17. Unwilling or unable to complete subject diary
18. Any other clinical condition, psychiatric condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable or to comply with follow-up visits

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Joslyn, Ph.D., Study Director — Sponsor GmbH
Locations (50):
- United States (27):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Helen F. Graham Cancer Center, Newark, Delaware
  - UF Health Cancer Center, Orlando, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - St. Vincent Anderson Regional, Cancer Center, Anderson, Indiana
  - Norton Cancer Institute, Multicisciplinary Clinic, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada-Henderson, Henderson, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Northwell Health Cancer Institute / Center for Novel Cancer Therapeutics, Lake Success, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, Albert Einstein College of Medicine, Department of Radiation Oncology, The Bronx, New York
  - Caromont Regional Medical Center, Gastonia, North Carolina
  - East Carolina Univ School of Dental Medicine, Greenville, North Carolina
  - Mercy Medical Center, Canton, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Temple University Hospital, Radiation Oncology, Philadelphia, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Radiation Oncology Moser, Charlottesville, Virginia
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Multicare Health Center, Gig Harbor, Washington
  - Cancer Care NW, Spokane, Washington
- Belgium (5):
  - Jules Bordet Institute, Brussels
  - University Hospital Brussels, Brussels
  - University Hospital Antwerp, Edegem
  - University Hospitals Leuven, Leuven
  - St. Maarten General Hospital, Mechelen
- Germany (13):
  - University Hospital Aachen, Aachen
  - Amper Hospital, Dachau
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Giessen and Marburg, Giessen
  - Hospital Kassel, Kassel
  - University Hospital Schleswig-Holstein, Kiel
  - Helios Hospital Krefeld, Krefeld
  - University Hospital Johannes Gutenberg - University of Mainz, Mainz
  - University Hospital Mannheim, Mannheim
  - Clinics Maria Hilf - Hospital St. Franziskus, Mönchengladbach
  - Ludwig Maximilians University Hospital, Munich
  - University Hospital Regensburg, Regensburg
  - Caritas Klinikum, Saarbrücken
- United Kingdom (5):
  - Derriford Hospital, Plymouth, Devon
  - Beatson West of Scotland Cancer Center, Glasgow
  - Guy's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Limaye SA, Haddad RI, Cilli F, Sonis ST, Colevas AD, Brennan MT, Hu KS, Murphy BA. Phase 1b, multicenter, single blinded, placebo-controlled, sequential dose escalation study to assess the safety and tolerability of topically applied AG013 in subjects with locally advanced head and neck cancer receiving induction chemotherapy. Cancer. 2013 Dec 15;119(24):4268-76. doi: 10.1002/cncr.28365. Epub 2013 Sep 24. PMID 24114811
- [Derived] Alexander LM, van Pijkeren JP. Modes of therapeutic delivery in synthetic microbiology. Trends Microbiol. 2023 Feb;31(2):197-211. doi: 10.1016/j.tim.2022.09.003. Epub 2022 Oct 8. PMID 36220750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients were randomized but never received study drug and are excluded from the safety analysis set.
Groups:
- AG013: Three rinses per day with AG013 mouth rinse beginning from the start of radiotherapy until 2 weeks following its completion for 7 to 9 weeks, depending on the duration of radiotherapy.
- Placebo: Three rinses per day with placebo mouth rinse beginning from the start of radiotherapy until 2 weeks following its completion for 7 to 9 weeks, depending on the duration of radiotherapy.
Period: Overall Study
Arm/Group | AG013 | Placebo
Started | 100 | 100
Completed | 67 | 60
Not Completed | 33 | 40
Not completed — Adverse Event | 4 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 12 | 27
Not completed — Symptomatic deterioration | 0 | 1
Not completed — Non-compliance | 2 | 0
Not completed — Other | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AG013 | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.98) | 60.4 (9.10) | 60.4 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 81 | 84 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 91 | 81 | 172
  Unknown or Not Reported | 7 | 12 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 93 | 92 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130
  Europe | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of AG013 Compared to Placebo for Reducing OM as Measured by Duration (in Days) of Severe Oral Mucositis (WHO Grades 3 or 4)
Description: Duration (in Days) of Severe Oral Mucositis (WHO Grades 3 or 4)
Time Frame: From the start of radiation therapy (RT) until 2 weeks following its completion, 7 to 9 weeks depending on the duration of CRT.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AG013 | Placebo
Number analyzed (Participants) | 100 | 100
Days
  US | 19.6 (25.00) | 20.6 (25.20)
  Europe | 17.2 (22.67) | 15.3 (22.54)

ADVERSE EVENTS:
Time Frame: From the time of screening and up to a total of 15 to 17 weeks, depending on the duration of CRT.
Description: Safety analyses were performed on the Safety Population which is comprised of all patients randomized to treatment and who received at least one dose of study drug.
  3 patients were randomized but never received study drug and are excluded from these analyses.
Arm/Group | AG013 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/100 | 4/97
Serious Adverse Events (participants affected / at risk) | 43/100 | 25/97
Other Adverse Events (participants affected / at risk) | 98/100 | 95/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG013 (N=100) | Placebo (N=97)
Nausea (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 6 | 4
Dysphagia (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 0
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Tracheostomy infection (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 3 | 4
General physical health deterioriation (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Administration site extravasation (General disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharynggeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiratoin (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AG013 (N=100) | Placebo (N=97)
Nausea (Gastrointestinal disorders) | 67 | 69
Constipation (Gastrointestinal disorders) | 54 | 41
Dry mouth (Gastrointestinal disorders) | 39 | 42
Vomiting (Gastrointestinal disorders) | 38 | 38
Dysphagia (Gastrointestinal disorders) | 33 | 39
Diarrhoea (Gastrointestinal disorders) | 27 | 43
Oral pain (Gastrointestinal disorders) | 17 | 14
Dyspepsia (Gastrointestinal disorders) | 15 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 5
Odynophagia (Gastrointestinal disorders) | 7 | 9
Saliva altered (Gastrointestinal disorders) | 8 | 4
Weight decreased (Investigations) | 29 | 29
White blood cell count decreased (Investigations) | 12 | 15
Blood creatinine increased (Investigations) | 14 | 10
Platelet count decreased (Investigations) | 10 | 12
Neutrophil count decreased (Investigations) | 11 | 10
Lymphocyte count decreased (Investigations) | 5 | 7
Alanine aminotransferase increased (Investigations) | 4 | 6
Blood urea increased (Investigations) | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 36 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 20 | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Fatigue (General disorders) | 56 | 58
Pyrexia (General disorders) | 14 | 9
Secretion discharge (General disorders) | 13 | 8
Asthenia (General disorders) | 5 | 4
Pain (General disorders) | 5 | 4
Localised oedema (General disorders) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 27 | 25
Dehydration (Metabolism and nutrition disorders) | 19 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 10
Malnutrition (Metabolism and nutrition disorders) | 7 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 5
Dysgeusia (Nervous system disorders) | 43 | 49
Headache (Nervous system disorders) | 24 | 21
Dizziness (Nervous system disorders) | 12 | 12
Candida infection (Infections and infestations) | 17 | 13
Oral candidiasis (Infections and infestations) | 20 | 6
Mucosal infection (Infections and infestations) | 6 | 8
Anaemia (Blood and lymphatic system disorders) | 21 | 33
Leukopenia (Blood and lymphatic system disorders) | 12 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 6
Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 6
Radiation skin injury (Injury, poisoning and procedural complications) | 32 | 45
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 2 | 5
Erythema (Skin and subcutaneous tissue disorders) | 15 | 9
Rash (Skin and subcutaneous tissue disorders) | 6 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 11 | 11
Anxiety (Psychiatric disorders) | 9 | 9
Tinnitus (Ear and labyrinth disorders) | 20 | 18
Ear pain (Ear and labyrinth disorders) | 6 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Hypotension (Vascular disorders) | 7 | 6
Acute kidney injury (Renal and urinary disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03234465/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03234465/SAP_001.pdf